CLINICAL TRIAL: NCT07322770
Title: Retrospective Evaluation of the Long-term Effectiveness of the CR500™ SINGLE-DOSE GEL Medical Device in Patients With Knee Osteoarthritis (KOA) Enrolled in the Clinical Study CTD-SW CR500™-KOA 2020
Brief Title: Retrospective Evaluation of the Long-term Effectiveness of the CR500™ SINGLE-DOSE GEL Medical Device in Patients With Knee Osteoarthritis (KOA)
Status: Completed | Type: Observational
Sponsor: Contrad Swiss SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CTD-SW CR500™-KOA 2020 - FU 25
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic Acid; Algofunctional Scores; Peptides; Knee Osteoarthritis; Topical Treatment; Patient Satisfaction
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CR500 single-dose gel: This retrospective phone follow-up involves the 35 patients who completed the CTD-SW CR500™-KOA 2020 study. After obtaining consent, patients will be asked whether and when they required further therapeutic interventions for KOA after the trial. This information will describe the long-term course of each arm by identifying subsequent treatments needed beyond the interventions originally administered during the study.
  Interventions: Device: CR 500™ SINGLE-DOSE GEL

INTERVENTIONS:
Device: CR 500™ SINGLE-DOSE GEL — CR 500™ SINGLE-DOSE GEL is a hydrogel to be applied to intact skin, useful to attenuate the physiological degeneration of cartilage typical of osteoarthritic processes. The presence of sodium hyaluronate facilitates the movement of joints and tendons for greater mobility and flexibility

SUMMARY:
Evaluate the long-term efficacy of the CR500™ therapy in patients with knee OA.

DETAILED DESCRIPTION:
To assess whether and when the patients enrolled in the CTD-SW CR500™-KOA 2020 clinical study required new orthopaedic treatment for knee osteoarthritis, starting at least 24 months after the conclusion of the clinical study.

Evaluate whether, in the long term, despite the potential bias of other therapies, treatment with CR500 has led to a lasting improvement, especially in comparison with infiltrative treatments based on the literature.

Collect data on patient satisfaction with the therapy received

ELIGIBILITY:
Inclusion Criteria:

* Oral informed consent from the patient.
* Participation in the CTD-SW CR500™-KOA 2020 clinical study.
* Willingness to participate in the survey.

Exclusion Criteria:

* Patients who were excluded following major protocol violations during the CTD-SW CR500™-KOA 2020 clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the CTD-SW CR500™-KOA 2020 clinical study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Lequesne Knee Index (LKI) Score | At least after 24 Months from the end of NCT05661162 study visit
  The primary efficacy endpoint of the study will be the evaluation of the long-term clinical performance of the CR500™, used as intended in patients affected by KOA, in variation of symptoms related to the physiological degeneration of cartilage typical of osteoarthritic processes, in terms of difference in LKI score between the end of NCT05661162 study visit and follow-up visit.
  Lequesne Knee Index Score:
  minimum index score: 0 maximum index score: 24
  0 means none OA
  >= means extremely severe OA

SECONDARY OUTCOMES:
Need for additional therapies before and after CR500™. | At least after 24 Months from the end of NCT05661162 study visit.
  To collect information, via a questionnaire, on the need for joint injections before and after CR500™ therapy.
  Did the patients receive HA infiltration before the therapy with CR500? Yes No
  Had the patients received another treatment for the same pathology after CR500™? Yes No
Timing and type of other interventions performed on the same knee with KOA treated with CR500™ in the NCT05661162 study. | At least after 24 Months from the end of NCT05661162 study visit
  To collect, via a questionnaire, information on the timing and type of other interventions performed on the same KOA-affected knee treated with CR500™ in the NCT05661162 study, as follows:
  After the treatment with CR500 have you undergone any other therapies for the treatment of OA? Yes No
  If yes, which ones? Infiltrative Therapies (HA, PRP, or corticosteroids) Oral anti-inflammatory or pain-relief therapies Topical anti-inflammatory or pain-relief therapies Electromedical therapies Physiotherapy
  Do you roughly remember when (month/year)?
Long-term satisfaction with the CR500™ treatment. | At least after 24 Months from the end of NCT05661162 study visit
  To collect, via a questionnaire, information on long-term patient satisfaction at least 24 months after the last application of CR500™.
  Would you repeat the treatment with CR500™? Yes No Uncertain
Recurrence of pain in the CR500™-treated knee and prosthesis status. | At least after 24 Months from the end of NCT05661162 study visit
  To collect, via a questionnaire, information on the health status of the knee treated with CR500™ (presence of pain after treatment) and on prosthesis status (whether undergone or scheduled).
  After the treatment with CR500, has a similar pain reappeared in the same knee? Yes Yes, but less intense No
  After the treatment with CR500, have you undergone knee replacement surgery? Yes Waiting list No If Yes, when?

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Mater Domini Casa di Cura Privata - Gruppo Humanitas, Castellanza, VARESE, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Colombini A, Doro G, Ragni E, Forte L, de Girolamo L, Zerbinati F. Treatment with CR500(R) improves algofunctional scores in patients with knee osteoarthritis: a post-market confirmatory interventional, single arm clinical investigation. BMC Musculoskelet Disord. 2023 Aug 12;24(1):647. doi: 10.1186/s12891-023-06754-7. PMID 37573322